CLINICAL TRIAL: NCT05422924
Title: A Pilot and Feasibility Study of a Web-based Platform to Improve Physical Function, Nutrition, and Mindfulness in Patients With Long COVID
Brief Title: A Web-based Platform to Improve Physical Function, Nutrition, and Mindfulness in Patients With Long COVID
Acronym: BLEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Revive Wellness Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00120894
Record Dates: First submitted 2022-06-16; First posted 2022-06-21 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Long COVID
Keywords: Nutrition; Physical activity; Feasibility; Body composition
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): No use of My Viva Plan
- Intervention Arm (Experimental): Use of My Viva Plan
  Interventions: Behavioral: Web-based platform. (My Viva Plan)

INTERVENTIONS:
Behavioral: Web-based platform. (My Viva Plan) — Participants will use a web-based platform (i.e. My Viva Plan®) to improve physical function, nutrition and mindfulness.
  Arms: Intervention Arm

SUMMARY:
Patients with COVID-19 may experience prolonged physical and psychological symptoms after weeks or months of the infection. This may be caused by a combination of factors including poor nutrition, low physical activity, and lack of emotional support. Leading to poor overall health and low quality of life. This evidence indicated that people with long COVID-19 need a personalized intervention. Our objective is to determine if the use of an online application that is based on preventive self-care and that includes nutrition and mindfulness will be feasible to use for patients with long COVID.

DETAILED DESCRIPTION:
A Canadian web-based platform called My Viva Plan® became available. This web-based platform is based on preventive self-care and it includes three key pillars of health: nutrition and mindfulness.

Long COVID patients will be randomized into the following two groups; intervention arm (will use a web-based platform for 8 weeks) vs. control arm (will not use a web-based platform for 8 weeks).The primary aim of this study is to investigate the feasibility (defined by recruitment, adherence, and retention) of an 8-week digital nutrition and mindfulness self-care intervention program using My Viva Plan® versus usual care (i.e. general advice) in patients with long COVID who continue to have signs and symptoms not explainable by other causes. Dietary intake, physical function, body composition and mental health variables will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years.
* COVID diagnosed (PCR positivity) >12 weeks at time of screening and have persistent symptoms.
* Body mass index (BMI) >18.5kg/m2 and < 35 kg/m2.
* People with long COVID syndrome diagnosis enrolled in the Kaye Edmonton Clinic.
* Have mild to moderate long COVID syndrome (Based on the Post COVID-19 Functional Status Scale from 0-3).

Exclusion Criteria:

* Patients with severe mobility impairment (People without sufficiently mobile to come to the study centre).
* Diagnosis of severe mental health disorders (e.g., depression, anxiety, eating disorders).
* Individuals with pacemakers or other internal electrical medical devices.
* Suffer from claustrophobia.
* Pregnancy or lactation.
* No internet access.
* Not able to understand and communicate in English.
* Major visual or hearing impairment or other serious illness that would preclude participation.
* Living in assisted living situations or a nursing home.
* Individuals who fell more than 3 times in the last month. Because of the risk of doing a physical activity unsupervised.
* Not willing to make a change in their lifestyle (Readiness to change).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility (defined by recruitment, adherence, and retention). | Baseline, week 8
  The proportion of participants that agreed to participate, the engagement in the platform (login), participants who complete both visits

SECONDARY OUTCOMES:
Changes in quality of life parameters | Baseline, week 8
  Changes in scores of quality of life assessed by EuroQol 5-level EQ-5D.
Changes in fat mass | Baseline, week 8
  Changes in fat mass (kg) using bioelectrical impedance analysis
Changes in lean mass | Baseline, week 8
  Changes in lean mass (kg) using bioelectrical impedance analysis
Changes in muscle cross sectional area | Baseline, week 8
  Changes in muscle cross sectional area (cm2) using an ultrasound
Changes in dietary intake | Baseline, week 8
  Changes in diet quality assessed by dietary intake assessed by Automated Self-Administered 24-hour dietary assessment tool and analysed with Canadian version of the Healthy Eating Index
Changes in mindfulness with Mental health questionnaire from the Symptom Burden Questionnaire for Long COVID | Baseline, week 8
  Changes in mindfulness assessed by Mental health questionnaire from the Symptom Burden Questionnaire for Long COVID (SBQ-LC). 9-item measure. Scores are to 0-100 linear. Higher scores indicate greater symptom burden.
Changes in self-efficacy assessed with Patient-Reported Outcomes Measurement Information System | Baseline, week 8
  Changes in self-efficacy for managing chronic conditions with of 8-item questionnaire that is based on a Patient-Reported Outcomes Measurement Information System (PROMIS).The total raw score (ranging from 8 to 40) will be transferred to a T-score. A mean of 50 and a standard deviation (SD) of 10 will be the average. A higher PROMIS T-score indicates that the respondent has greater self-efficacy for managing their emotions than the general chronic condition population.
Changes in physical function | Baseline, week 8
  Changes in physical function assessed by handgrip strength
Changes in physical performance | Baseline, week 8
  Changes in physical performance assessed by 6-minute walk test
Changes in physical activity (daily activities subscale) by the Symptom Burden Questionnaire for Long COVID. | Baseline, week 8
  Changes in physical activity assessed by Daily Activities Symptom Burden Questionnaire for Long COVID (SBQ-LC). Raw scores (ranging from 0 to 24) will be converted to 0-100 linear scores with conversion tables. Higher scores indicate greater symptom burden.
Changes in physical activity using the International Physical Activity Questionnaire | Baseline, week 8
  Changes in physical activity assessed by International Physical Activity Questionnaire (IPAQ). This questionnaire collects information about three specific types of physical activity: walking, moderate-intensity activities and vigorous intensity activities. To compute the total score, measures of frequency (measured in days per week) and duration (time per day) are needed. We will use this information to compare over time.
Changes in resting energy expenditure | Baseline, week 8
  Changes in resting energy expenditure assessed by a metabolic cart (indirect calorimetry)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Prado, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No